CLINICAL TRIAL: NCT00554515
Title: The High-Dose Aldesleukin (IL-2) "Select" Trial: A Trial Designed to Prospectively Validate Predictive Models of Response to High Dose IL-2 Treatment in Patients With Metastatic Renal Cell Carcinoma
Brief Title: The High-Dose Aldesleukin (IL-2) "Select" Trial for Patients With Metastatic Renal Cell Carcinoma
Acronym: SELECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: City of Hope National Medical Center (Other); Providence Cancer Center, Earle A. Chiles Research Institute (Other); Dartmouth-Hitchcock Medical Center (Other); Indiana University (Other); Loyola University (Other); Our Lady of Mercy Medical Center (Other); Roswell Park Cancer Institute (Other); University of California, Los Angeles (Other); University of Cincinnati (Other); University of Pittsburgh (Other); University of Virginia (Other); Vanderbilt University (Other); Wayne State University (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, David McDermott, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFHCC 06-149; NCT00536757 (obsolete NCT alias)
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Kidney; Renal Cell; Metastatic; interleukin-2; select
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HD IL2 (Experimental): Participants received high-dose (HD) IL2, 600,000 IU/kg/dose (Prometheus Laboratories Inc.) i.v. every 8 hours for 5 days (maximum of 14 doses) beginning on day 1 and again on day 15. One course generally consisted of 5 days of treatment, 9 days of rest, 5 more days of treatment, and 9 weeks of rest, followed by up to two additional courses of HD IL2 for patients who benefited and tolerated most of the planned IL2 doses. A treatment delay of up to 4 weeks was allowed for resolution of side effects between courses. Patients were eligible to receive a maximum of three courses of treatment.
  Interventions: Drug: HD IL2

INTERVENTIONS:
Drug: HD IL2
  Other Names: Proleukin; Aldesleukin

SUMMARY:
High-dose interleukin 2 (Proleukin, Novartis) (IL-2) is approved by the U.S Food and Drug Administration (FDA) for the treatment of metastatic kidney cancer and is a standard treatment of this disease. At the present time, IL-2 is the only therapy for kidney cancer that can produce a remission of disease that lasts after treatment is completed. However, most patients who receive IL-2 do not benefit and all patients experience potentially dangerous side effects.

Recent research has suggested that certain patients may respond better to IL-2 than others. The Cytokine Working Group is currently conducting a clinical trial that aims to identify and confirm this research and narrow the application of IL-2 to those patients most likely to benefit.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine, in a prospective fashion, if the response rate to high-dose IL-2 for patients with metastatic renal cell carcinoma and "good" pathologic predictive features is significantly higher than a historical, unselected patient population.

Secondary

* To determine, in a prospective fashion, the response rate to high-dose IL-2 for patients with metastatic renal cell carcinoma and "poor" pathologic predictive features and to compare this response rate to the response rate of patients with "good" pathologic predictive features.
* To determine if components of other predictive and prognostic models (e.g MSKCI or UCLA criteria) can help to further define the optimal population to receive high-dose IL2 for metastatic renal cell carcinoma.
* To identify features of the baseline immune function (arginine, arginase, T cell zeta chain) of patients with metastatic renal cell carcinoma that are associated with response to high-dose IL-2.
* To identify new proteins or patterns of gene expression that might be associated with high-dose IL-2 responsiveness in order to further narrow the application of IL-2 therapy to those who will benefit the most.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed renal cell carcinoma that is metastatic or unresectable.
* If patients have measurable disease restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology.
* Patients must provide access to tissue blocks containing adequate tumor for interpretation and analysis.
* Patients must have measurable disease.
* Patients must have good performance status (ECOG 0 or 1; Karnofsky PS 100-80%).
* Patients must have adequate organ function.
* Patients must have no contraindication of vasopressor agents.
* Patients must be ≥ 18 years of age.

Exclusion Criteria:

* Patients who have received systemic therapy for metastatic disease.
* Patients with organ allografts.
* Patients who require or are likely to require systemic corticosteroid therapy for intercurrent illness.
* Patients with any significant medical disease other than the malignancy (e.g. COPD, patients with ascites or pleural effusions), which in the opinion of the investigator would significantly increase the risk of immunotherapy.
* Patients with a history of another malignancy within the past 5 years other than surgically cured non-melanoma skin cancer, carcinoma-in-situ or Stage I carcinoma of the cervix.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2006-11; Primary Completion 2013-10-31 (Actual); Study Completion 2013-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F McDermott, MD, Study Chair — Beth Israel Deaconess Medical Center; Kim Margolin, MD, Principal Investigator — City of Hope National Medical Center; Walter Urba, MD, Principal Investigator — Chiles Cancer Center; Marc Ernstoff, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Theodore Logan, MD, Principal Investigator — Indiana University; Joseph Clark, MD, Principal Investigator — Loyola University; Janice Dutcher, MD, Principal Investigator — Our Lady of Mercy Cancer Center; Michael Wong, MD, Principal Investigator — Roswell Park Cancer Institute; Allen Pantuck, MD, Principal Investigator — University of California, Los Angeles; Leslie Oleksowicz, MD, Principal Investigator — University of Cincinnati; Leonard Appleman, MD, Principal Investigator — University of Pittsburgh; Geoffrey Weiss, MD, Principal Investigator — University of Virginia; Jeffrey Sosman, MD, Principal Investigator — Vanderbilt University; Ulka Vaishampayan, MD, Principal Investigator — Wayne State University
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDermott DF. Update on the application of interleukin-2 in the treatment of renal cell carcinoma. Clin Cancer Res. 2007 Jan 15;13(2 Pt 2):716s-720s. doi: 10.1158/1078-0432.CCR-06-1872. PMID 17255299 (Retraction: PMID 30087149 Clin Cancer Res. 2018 Aug 1;24(15):3783)
- [Background] Atkins M, Regan M, McDermott D, Mier J, Stanbridge E, Youmans A, Febbo P, Upton M, Lechpammer M, Signoretti S. Carbonic anhydrase IX expression predicts outcome of interleukin 2 therapy for renal cancer. Clin Cancer Res. 2005 May 15;11(10):3714-21. doi: 10.1158/1078-0432.CCR-04-2019. PMID 15897568
- [Result] McDermott DF, Cheng SC, Signoretti S, Margolin KA, Clark JI, Sosman JA, Dutcher JP, Logan TF, Curti BD, Ernstoff MS, Appleman L, Wong MK, Khushalani NI, Oleksowicz L, Vaishampayan UN, Mier JW, Panka DJ, Bhatt RS, Bailey AS, Leibovich BC, Kwon ED, Kabbinavar FF, Belldegrun AS, Figlin RA, Pantuck AJ, Regan MM, Atkins MB. The high-dose aldesleukin "select" trial: a trial to prospectively validate predictive models of response to treatment in patients with metastatic renal cell carcinoma. Clin Cancer Res. 2015 Feb 1;21(3):561-8. doi: 10.1158/1078-0432.CCR-14-1520. Epub 2014 Nov 25. PMID 25424850

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from 13 institutions between November 2006 and November 2008.
Period: Overall Study
Arm/Group | HD IL2
Started | 123
Treated (3 participants withdrew consent before starting treatment.) | 120
Completed | 5
Not Completed | 118
Not completed — Withdrawal by Subject | 3
Not completed — Disease progression | 52
Not completed — Physician Decision | 18
Not completed — Withdrawal by Subject | 11
Not completed — Adverse Event | 9
Not completed — Death | 2
Not completed — Achieved Stable Disease | 7
Not completed — Other | 1
Not completed — Misc | 15

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated participants.
Arm/Group | HD IL2
Number analyzed (Participants) | 120
Age, Continuous [Median (Full Range); unit: years] | 56 [28 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 85
Region of Enrollment [Number; unit: participants]
  United States | 120
MSKCC Risk Group [Count of Participants; unit: Participants] — Memorial Sloan Kettering Cancer Center (MSKCC) Risk Group: MSKCC developed a nomogram that is used to classify patients into 3 renal cell carcinoma (RCC) 5-year disease recurrence risk groups (low, intermediate, and high) using data from patients treated at MSKCC. The components of the nomogram include RCC histology, disease symptoms, pT stage, and tumor size.
  Participants
    Favorable | 23
    Intermediate | 84
    Poor | 13
UCLA SANI Score [Count of Participants; unit: Participants] — University of California Los Angeles (UCLA) Survival After Nephrectomy and Immunotherapy (SANI) score: This tool also predicts RCC patient's survival based on lymph node status, metastases, sarcomatoid feature, and TSH level. Patients are classified into 3 groups (low, intermediate, and high). [Leibovich et al. Cancer 2003]
  Participants
    Low | 10
    Intermediate | 102
    High | 8
ISM Risk Group [Count of Participants; unit: Participants] — ISM [Atkins et al CCR 2005] Pathology [Upton et al. J Immunother 2005] CAIX (carbonic anhydrase IX) [Bui et al. CCR 2003]
  Poor: Poor predictive pathology OR the combination of intermediate predictive pathology and low CAIX staining Good: Good predictive pathology OR the combination of intermediate predictive pathology and high CAIX staining
  Participants
    Good | 74
    Poor | 43
    Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response in ISM Good Risk Group
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) on treatment based on World Health Organization (WHO) criteria. [Miller et al. Cancer 1981] Per WHO, evaluation of tumor measurements of measurable lesions centers on the percent change from baseline in the sum of the perpendicular diameters. Complete Response (CR) is disappearance of all clinical and laboratory evidence of disease; Partial Response (PR) is a >/= 50% decrease. PR status also requires no simultaneous increase in the size of any metastatic lesion, absence of one or more new metastatic lesions and/or unequivocal progression of existing non-target lesions. CR and PR status needs confirmation within 4 weeks. Response status was determined by investigator assessment of radiographs.
Time Frame: Disease was evaluated radiologically at baseline and during weeks 8 and 12 of each course. Participants received up to 3 courses of 12 weeks duration each. Median (range) days on treatment: 20 (1-262).
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data for ISM analysis and classified as ISM good risk.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- ISM Good Risk Group: ISM [Atkins et al CCR 2005]:
  Good predictive pathology OR the combination of intermediate predictive pathology and high CAIX staining
  Pathology [Upton et al. J Immunother 2005] Good predictive pathology: clear-cell histology AND no papillary features AND >50% alveolar features AND no granular features Intermediate predictive pathology: clear-cell histology AND no papillary features AND some (>0%) alveolar features AND 50% granular features
  CAIX [Bui et al. CCR 2003] High CAIX staining: >85% of CAIX positive tumor cells
Arm/Group | ISM Good Risk Group
Number analyzed (Participants) | 74
proportion of participants | .23 [.14 to .34]
Statistical Analysis 1: Comparison: ISM Good Risk Group; Test type: Superiority — Comparison against historical control ORR of 14%; p = 0.042, exact binomial test

2. Secondary Outcome: Objective Response Rate in ISM Poor Risk Group
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on treatment on World Health Organization (WHO) criteria. [Miller et al. Cancer 1981] Per WHO, evaluation of tumor measurements of measurable lesions centers on the percent change from baseline in the sum of the perpendicular diameters. Complete Response (CR) is disappearance of all clinical and laboratory evidence of disease; Partial Response (PR) is a >/= 50% decrease. PR status also requires no simultaneous increase in the size of any metastatic lesion, absence of one or more new metastatic lesions and/or unequivocal progression of existing non-target lesions. CR and PR status needs confirmation within 4 weeks. Response status was determined by independent assessment of radiographs.
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data for ISM analysis and classified as ISM poor risk.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- ISM Poor Risk Group: ISM [Atkins et al CCR 2005]:
  Poor predictive pathology OR the combination of intermediate predictive pathology and low CAIX staining
  Pathology [Upton et al. J Immunother 2005] Poor predictive pathology: non-clear-cell histology OR some (>0%) papillary features OR no alveolar features OR >50% granular features Intermediate predictive pathology: clear-cell histology AND no papillary features AND some (>0%) alveolar features AND 50% granular features
  CAIX [Bui et al. CCR 2003] Low CAIX staining: </=85% of CAIX positive tumor cells
Arm/Group | ISM Poor Risk Group
Number analyzed (Participants) | 43
proportion of participants | .23 [.14 to .34]
Statistical Analysis 1: Comparison: ISM Poor Risk Group; Objective response rates were compared between ISM good and poor risk subgroups. ISM good risk ORR reported under primary endpoint; Test type: Superiority; p = 0.39, Fisher Exact

3. Secondary Outcome: Objective Response Rate (Independent Assessment)
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) on treatment based on World Health Organization (WHO) criteria. [Miller et al. Cancer 1981] Per WHO, evaluation of tumor measurements of measurable lesions centers on the percent change from baseline in the sum of the perpendicular diameters. Complete Response (CR) is disappearance of all clinical and laboratory evidence of disease; Partial Response (PR) is a >/= 50% decrease. PR status also requires no simultaneous increase in the size of any metastatic lesion, absence of one or more new metastatic lesions and/or unequivocal progression of existing non-target lesions. CR and PR status needs confirmation within 4 weeks.. Response status was determined by independent assessment of radiographs.
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | HD IL2
Number analyzed (Participants) | 120
proportion of participants | .25 [.175 to .337]
Statistical Analysis 1: Comparison: HD IL2; Test against the historical ORR was conducted in the overall study population as secondary analyses; Test type: Superiority; p = 0.0014, exact binomial test

4. Secondary Outcome: Overall Survival
Description: Overall survival based on the Kaplan-Meier method is defined as the time from treatment start to date of death or censored at the date of last documented contact.
Time Frame: Participants were followed for survival up to 7 years.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HD IL2
Number analyzed (Participants) | 120
months | 42.8 [35.6 to 51.9]

5. Secondary Outcome: 3-Year Progression-Free Survival Rate
Description: 3-year progression-free survival rate is defined as the proportion of patients absent death or progression based on WHO criteria by 3 years since time of treatment start. PD is a >/=25% increase in the sum of products of the perpendicular diameters of all measurable lesions. Further, PD is the appearance of one or more new metastatic lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and during weeks 8 and 12 of each course. Long-term follow-up occurred every 3 m for 2 yrs, semi-annually for yr 3 and annually for yrs 4 and 5. Relevant for this endpoint was disease status at 3 y.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | HD IL2
Number analyzed (Participants) | 120
proportion of participants | .108 [.065 to .167]

6. Secondary Outcome: Objective Response Rate by MSKCC Risk Group
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) on treatment based on World Health Organization (WHO) criteria. [Miller et al. Cancer 1981] Per WHO, evaluation of tumor measurements of measurable lesions centers on the percent change from baseline in the sum of the perpendicular diameters. Complete Response (CR) is disappearance of all clinical and laboratory evidence of disease; Partial Response (PR) is a >/= 50% decrease. PR status also requires no simultaneous increase in the size of any metastatic lesion, absence of one or more new metastatic lesions and/or unequivocal progression of existing non-target lesions. CR and PR status needs confirmation within 4 weeks. Response status was determined by independent assessment of radiographs.
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Favorable MSKCC Risk Group; Intermediate MSKCC Risk Group; Poor MSKCC Risk Group: MSKCC developed a nomogram that is used to classify patients into 3 renal cell carcinoma (RCC) 5-year disease recurrence risk groups (low, intermediate, and high) using data from patients treated at MSK. The components of the nomogram include RCC histology, disease symptoms, pT stage, and tumor size.
Arm/Group | Favorable MSKCC Risk Group | Intermediate MSKCC Risk Group | Poor MSKCC Risk Group
Number analyzed (Participants) | 23 | 84 | 13
proportion of participants | .22 [.07 to .44] | .25 [.16 to .36] | .31 [.09 to .61]
Statistical Analysis 1: Comparison: Favorable MSKCC Risk Group vs Intermediate MSKCC Risk Group vs Poor MSKCC Risk Group; Objective response rates were compared between MSKCC subgroups; Test type: Superiority; p = .89, Fisher Exact

7. Secondary Outcome: Objective Response Rate by UCLA SANI Score
Description: as for outcome 6
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Low UCLA SANI Score; Intermediate UCLA SANI Score; High UCLA SANI Score: This tool predicts RCC patient's survival based on lymph node status, metastases, sarcomatoid feature, and TSH level. Patients are classified into 3 groups (low, intermediate, and high).
Arm/Group | Low UCLA SANI Score | Intermediate UCLA SANI Score | High UCLA SANI Score
Number analyzed (Participants) | 10 | 102 | 8
proportion of participants | .20 [.03 to .56] | .27 [.19 to .37] | .00 [.00 to .37]

8. Secondary Outcome: Objective Response Rate by Tumor Type
Description: as for outcome 6
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Clear Cell Tumor Type | Non-clear Cell Tumor Type
Number analyzed (Participants) | 114 | 5
proportion of participants | .26 [.19 to .35] | .00 [0.00 to 0.52]
Statistical Analysis 1: Comparison: Clear Cell Tumor Type vs Non-clear Cell Tumor Type; Objective response rates were compared between tumor type subgroups; Test type: Superiority; p = .33, Fisher Exact

9. Secondary Outcome: Objective Response Rate by Clear Cell Histology Risk Group
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on World Health Organization (WHO) criteria. [Miller et al. Cancer 1981] Per WHO, evaluation of tumor measurements of measurable lesions centers on the percent change from baseline in the sum of the perpendicular diameters. Complete Response (CR) is disappearance of all clinical and laboratory evidence of disease; Partial Response (PR) is a >/= 50% decrease. PR status also requires no simultaneous increase in the size of any metastatic lesion, absence of one or more new metastatic lesions and/or unequivocal progression of existing non-target lesions. CR and PR status needs confirmation within 4 weeks.
Time Frame: Disease was evaluated radiologically at baseline and during weeks 8 and 12 of each course. Response status was confirmed by an independent assessment of radiographs. Participants received up to 3 courses of 12 weeks duration each.
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Good Clear Cell Histology Risk Group | Intermediate Clear Cell Histology Risk Group | Poor Clear Cell Histology Risk Group
Number analyzed (Participants) | 11 | 83 | 25
proportion of participants | .27 [.06 to .61] | .24 [.15 to .35] | .28 [.12 to .49]
Statistical Analysis 1: Comparison: Good Clear Cell Histology Risk Group vs Intermediate Clear Cell Histology Risk Group vs Poor Clear Cell Histology Risk Group; Objective response rates were compared between clear cell histology subgroups; Test type: Superiority; p = .89, Fisher Exact

10. Secondary Outcome: Objective Response Rate by CA-9 Score (CAIX Classification)
Description: as for outcome 6
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- High CA-9 Score: This score is based on the expression of the CA 9 protein (encoded by the CA9 gene) assessed from patient's tumor specimen. CA 9 expression score is quantified by immunohistochemical analysis using CA9 monoclonal antibody (M75); High is >85% of CAIX positive tumor cells.
- Low CA-9 Score: This score is based on the expression of the CA 9 protein (encoded by the CA9 gene) assessed from patient's tumor specimen. CA 9 expression score is quantified by immunohistochemical analysis using CA9 monoclonal antibody (M75); Low is </=85% of CAIX positive tumor cells
Arm/Group | High CA-9 Score | Low CA-9 Score
Number analyzed (Participants) | 78 | 39
proportion of participants | .33 [.19 to .50] | .22 [.13 to .33]
Statistical Analysis 1: Comparison: Low CA-9 Score; Objective response rates were compared between CA-9 score subgroups; Test type: Superiority; p = .19, Fisher Exact

11. Secondary Outcome: Objective Response Rate by PD-L1 Tumor
Description: as for outcome 6
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | PD-L1 Tumor Negative | PD-L1 Tumor Positive
Number analyzed (Participants) | 95 | 18
proportion of patients | .19 [.12 to .28] | .50 [.26 to .74]
Statistical Analysis 1: Comparison: PD-L1 Tumor Negative vs PD-L1 Tumor Positive; Objective response rates were compared between PD-L1 tumor subgroups; Test type: Superiority; p = 0.01, Fisher Exact

12. Secondary Outcome: Objective Response Rate by B7-H3 Tumor
Description: as for outcome 6
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Negative | Positive
Number analyzed (Participants) | 29 | 86
proportion of participants | .11 [.02 to .28] | .29 [.20 to .40]
Statistical Analysis 1: Comparison: Negative vs Positive; Objective response rates were compared between B7-H3 tumor subgroups; Test type: Superiority; p = .08, Fisher Exact

13. Secondary Outcome: Objective Response Rate by CA-9 SNP
Description: as for outcome 6
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients with available tumor tissue/data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- CA-9 SNP Homozygous; CA-9 SNP Variant: Patient's SNP (Single Nucleotide Polymorphism) status is determined by sequencing their tumor specimens. Patients are classified as homozygous or variant based on the observed nucleotide sequence.
Arm/Group | CA-9 SNP Homozygous | CA-9 SNP Variant
Number analyzed (Participants) | 66 | 12
proportion of participants | .20 [.11 to .31] | .33 [.10 to .65]
Statistical Analysis 1: Comparison: CA-9 SNP Homozygous vs CA-9 SNP Variant; Objective response rates were compared between CA-9 SNP subgroups; Test type: Superiority; p = .28, Fisher Exact

14. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from treatment start to date of disease progression (PD) or death. Per WHO criteria: PD is a >/=25% increase in the sum of products of the perpendicular diameters of all measurable lesions. Further, PD is the appearance of one or more new metastatic lesions and/or unequivocal progression of existing non-target lesions. Participants who were event-free were censored at the date of their last disease evaluation.
Time Frame: Disease was evaluated radiologically at baseline and during weeks 8 and 12 of each course. Long-term follow-up occurred every 3 m for 2 yrs, semi-annually for yr 3 and annually for yrs 4 and 5. Median survival follow-up was X months (95% CI: ).
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HD IL2
Number analyzed (Participants) | 120
months | 4.2 [2.5 to 4.7]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed continuously throughout treatment. Treatment duration was a median of 3 courses (duration of 12 weeks each) in this study cohort. Note: one grade 2 serious adverse event (SAE), one grade 3 other adverse event (OAE) and one grade 4 OAE are missing from the tables because codes/description of these events are unknown but these patients are included in the overall number affected.
Description: Serious AEs: AE that results in death; is life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly or birth defect; or is an important medical event when, based upon appropriate medical judgment, it may jeopardize the participant and require medical or surgical intervention to prevent one of the above outcomes. Other AEs: Remaining AEs (max grade) with trt-attribution of possibly, probably or definitely.
Arm/Group | HD IL2
All-Cause Mortality (participants affected / at risk) | 3/120
Serious Adverse Events (participants affected / at risk) | 15/120
Other Adverse Events (participants affected / at risk) | 2/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HD IL2 (N=120)
Hemoglobin (Blood and lymphatic system disorders) | 1
Cardiac-ischemia (Cardiac disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
Cardiac-other (Cardiac disorders) | 2
Fatigue (General disorders) | 3
Fever w/o neutropenia (General disorders) | 1
Constitutional, other (General disorders) | 1
Liver dysfunction/failure (Hepatobiliary disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Lymphopenia (Investigations) | 2
Platelets (Investigations) | 1
Bilirubin (Investigations) | 3
Creatinine (Investigations) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Confusion (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HD IL2 (N=120)
Renal failure (Renal and urinary disorders) | 1
Uveitis (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No